CLINICAL TRIAL: NCT02164357
Title: Efficacy and Security of an Endovascular Treatment as First Choice Procedure Compared With a Standard Intravenous Thrombolytic Therapy Treatment for Patients With Acute Ischemic Stroke Within 4.5 Hours After Onset: A Prospective Cohorts Study
Brief Title: Efficacy and Security of an Endovascular Treatment as First Choice Procedure Compared With a Standard Intravenous Thrombolytic Therapy Treatment for Patients With Acute Ischemic Stroke Within 4.5 Hours After Onset
Acronym: FUN-TPA
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Other Study IDs: FUN-TPA-2012-01
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-06

CONDITIONS: Acute Ischaemic Stroke
Keywords: Ischaemic Stroke; Main artery occlusion; Endovascular treatment; Intravenous Thrombolytic Therapy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- EVT: Patients receiving endovascular treatment (EVT) within 4.5 hours after onset because intravenous thrombolytic therapy (IVT) is contraindicated
  Interventions: Procedure: EVT (endovascular treatment )
- IVT + EVT: Patients receiving intravenous thrombolytic therapy (IVT) followed by endovascular treatment (EVT) within 4.5 hours after onset
  Interventions: Procedure: EVT (endovascular treatment ); Procedure: IVT (intravenous thrombolytic therapy)
- IVT (intravenous thrombolytic therapy): Patients that will received IVT only within 4.5 hours after onset
  Interventions: Procedure: IVT (intravenous thrombolytic therapy)

INTERVENTIONS:
Procedure: EVT (endovascular treatment )
  Groups: EVT; IVT + EVT
Procedure: IVT (intravenous thrombolytic therapy)
  Groups: IVT (intravenous thrombolytic therapy); IVT + EVT

SUMMARY:
This study will compare two ways of treatment for acute ischemic stroke: an endovascular treatment (EVT), defined as intraarterial thrombolysis and/or mechanical thrombectomy as a first choice treatment versus intravenous thrombolytic therapy (IVT) only or followed by EVT in patients with acute ischemic stroke due to a main brain artery occlusion within 4.5 hours after onset. Patients treated with IVT only or with IVT followed by EVT will be analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

* 80 or less years old patients with acute stroke produced by a main artery occlusion
* NIHSS National Institutes of Health Stroke Scale score greater than 6 (severe neurological impairment)
* Patients receiving EVT or IVT within 4.5 hours after onset

Exclusion Criteria:

* EVT or IVT contraindication
* Previous neurological impairment, severe concomitant disease or poor prognosis.
* Pregnancy or breastfeeding
* Known hypersensitivity to any study drugs
* Severe organic disease for which there is not risk compensation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients younger than 80 with acute ischemic stroke produced by a main artery oclussion with a NIHSS > 6 (National Institute of Health Stroke Scale) receiving IVT or EVT within 4.5 hours after onset.
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2012-09; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Death within 90 days after onset | 90 days
Symptomatic intracranial haemorrhage | 7 days

SECONDARY OUTCOMES:
Stroke recovery rate after discharge | From onset to discharge
  Recovery defined as a 10-fold decrease in NIHSS or NIHSS (7 days after onset or at discharge)
Functional recovery | 4.5 hours after onset
  Modified Rankin Score (RMS) value

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Doce de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid

REFERENCES:
- [Derived] Alonso de Lecinana M, Martinez-Sanchez P, Garcia-Pastor A, Kawiorski MM, Calleja P, Sanz-Cuesta BE, Diaz-Otero F, Frutos R, Sierra-Hidalgo F, Ruiz-Ares G, Fandino E, Diez-Tejedor E, Gil-Nunez A, Fuentes B. Mechanical thrombectomy in patients with medical contraindications for intravenous thrombolysis: a prospective observational study. J Neurointerv Surg. 2017 Nov;9(11):1041-1046. doi: 10.1136/neurintsurg-2016-012727. Epub 2016 Nov 7. PMID 27821473
- [Derived] Kawiorski MM, Martinez-Sanchez P, Garcia-Pastor A, Calleja P, Fuentes B, Sanz-Cuesta BE, Lourido D, Marin B, Diaz-Otero F, Vicente A, Sierra-Hidalgo F, Ruiz-Ares G, Diez-Tejedor E, Fandino E, Alonso de Lecinana M. Alberta Stroke Program Early CT Score applied to CT angiography source images is a strong predictor of futile recanalization in acute ischemic stroke. Neuroradiology. 2016 May;58(5):487-93. doi: 10.1007/s00234-016-1652-7. Epub 2016 Feb 2. PMID 26838587